CLINICAL TRIAL: NCT03443713
Title: Evaluation of Physician-based Decision Support in Patients With Type 1 Diabetes on Multiple Daily Injection Therapy
Brief Title: Evaluation of Physician-based Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Jessica Castle, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18023
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus; MDI; CGM; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects randomly assigned to one of three types of exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Aerobic exercise (Experimental): Subjects in this arm will complete aerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.
  Interventions: Device: Dexcom G6 CGM
- Anaerobic exercise (Experimental): Subjects in this arm will complete anaerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.
  Interventions: Device: Dexcom G6 CGM
- High intensity interval exercise (Experimental): Subjects in this arm will complete high intensity interval exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.
  Interventions: Device: Dexcom G6 CGM

INTERVENTIONS:
Device: Dexcom G6 CGM — Subjects will wear a Dexcom G6 CGM for the 28 days they are on study.

SUMMARY:
The goal of this study is to assess the impact of physician-driven insulin setting changes in type 1 patients using multiple daily injection insulin therapy with exercise. This is a short outpatient study with multiple outpatient and home exercise sessions with an assigned type of exercise.

DETAILED DESCRIPTION:
Subjects will be on study for 28 days. Sensor glucose, exercise, insulin and meal data will be collected during this time. Subjects will wear the Dexcom G6 CGM system and a physical activity monitor. The Subjects will complete 2 exercise visits in-clinic and 4 exercise visits as an outpatient. Subjects will be randomized to aerobic, anaerobic or high intensity interval exercise sessions for 30 minutes each. Physicians will review CGM and insulin data every 7 days and make insulin dose recommendations that the subject will adjust in the dose calculator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 18 to 50 years of age.
* Physically willing and able to perform 30 min of exercise (as determined by the investigator after reviewing the subject's activity level).
* Use of multiple daily insulin injections (MDI).
* A1C ≥7.0% at the time of screening.
* Current use of a smart phone.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
* Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as reported by the OHSU laboratory).
* Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
* Hematocrit of less than 36% for men, less than 32% for women.
* History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator. Subjects will complete a hypoglycemia awareness questionnaire. Subjects will be excluded for four or more R responses.
* Adrenal insufficiency.
* Any active infection.
* Known or suspected abuse of alcohol, narcotics, or illicit drugs.
* Seizure disorder.
* Active foot ulceration.
* Peripheral arterial disease.
* Major surgical operation within 30 days prior to screening.
* Use of an investigational drug within 30 days prior to screening.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Bleeding disorder or platelet count below 50,000.
* Allergy to aspart or glargine insulin.
* Need for uninterrupted treatment of acetaminophen.
* Current administration of oral or parenteral corticosteroids.
* Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
* Beta blockers or non-dihydropyridine calcium channel blockers.
* Current use of any medication intended to lower glucose other than insulin (ex. use of liraglutide).
* A positive response to any of the questions from the Physical Activity Readiness Questionnaire with one exception: subject will not be excluded if he/she takes a single blood pressure medication that doesn't impact heart rate and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg).
* Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
* Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Castle, MD, Principal Investigator — Oregon Health and Science University; Peter Jacobs, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tyler NS, Mosquera-Lopez CM, Wilson LM, Dodier RH, Branigan DL, Gabo VB, Guillot FH, Hilts WW, El Youssef J, Castle JR, Jacobs PG. An artificial intelligence decision support system for the management of type 1 diabetes. Nat Metab. 2020 Jul;2(7):612-619. doi: 10.1038/s42255-020-0212-y. Epub 2020 Jun 1. PMID 32694787

RESULTS

PARTICIPANT FLOW:
Period: Start up Visit (2 Hours)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 9
Completed | 8 | 8 | 9
Not Completed | 0 | 0 | 0
Period: First at Home Period (9-14 Days)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 9
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: First Exercise Visit (1 Hour)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Dexcom Insertion Visit (30 Minutes)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Second at Home Period (2-11 Days)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Second Exercise Visit (1 Hour)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Third at Home Period (8-12 Days)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Close-out Visit (30 Minutes)
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aerobic Exercise; Anaerobic Exercise; High Intensity Interval Exercise: All study subjects were randomized to either aerobic, anaerobic or high intensity interval training. Subjects were on study for 28 days.
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 25
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.7) | 28.6 (6.0) | 29 (5.3) | 29.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 15
  Male | 4 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 7 | 4 | 8 | 19
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time With Sensed Glucose 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using values uploaded to Dexcom Clarity. The percent of time with sensed glucose 70-180 mg/dl was averaged across days 1-7.
Time Frame: Days 1-7
Population: 25 subjects were enrolled. One subject assigned to High intensity interval exercise dropped out before completing the exercise visits.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Aerobic Exercise: Subjects in this arm will complete aerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.Subjects are on study for 28 days.
- Anaerobic Exercise: Subjects in this arm will complete anaerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.Subjects are on study for 28 days.
- High Intensity Interval Exercise: Subjects in this arm will complete high intensity interval exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM.Subjects are on study for 28 days.
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 58.8 (18.9) | 51.2 (10.8) | 59.3 (14.6)

2. Primary Outcome: Percent of Time With Sensed Glucose Less Than 70 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 70 mg/dl using values uploaded to Dexcom Clarity.The percent of time with sensed glucose less than 70 mg/dl was averaged across days 1-7.
Time Frame: Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Anaerobic Exercise: Subjects in this arm will complete anaerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM. Subjects are on study for 28 days.
- High Intensity Interval Exercise: Subjects in this arm will complete high intensity interval exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM. Subjects are on study for 28 days.
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 3.3 (3.5) | 2.4 (1.4) | 3.3 (2.2)

3. Primary Outcome: Percent of Time With Sensed Glucose 70-180 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values between 70-180 mg/dl using values uploaded to Dexcom Clarity.The percent of time with sensed glucose 70-180 mg/dl was averaged across days 22-28.
Time Frame: Days 22-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Aerobic Exercise: Subjects in this arm will complete aerobic exercise at home and at OHSU for the study. Subjects will use a Dexcom G6 CGM. Subjects are on study for 28 days.
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 53.6 (13.6) | 51.0 (16.0) | 50.4 (13.4)

4. Primary Outcome: Percent of Time With Sensed Glucose Less Than 70 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 70 mg/dl using values uploaded to Dexcom Clarity.The percent of time with sensed glucose less then 70 mg/dl was averaged across days 22-28.
Time Frame: Days 22-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 3.8 (3.4) | 2.2 (2.4) | 3.1 (4.0)

5. Secondary Outcome: Percent of Time With Sensed Glucose Less Than 54 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 54 mg/dl using values uploaded to Dexcom Clarity.The percent of time with sensed glucose less then 54 mg/dl was averaged across days 1-7.
Time Frame: Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 0.5 (0.8) | 0.4 (0.3) | 0.5 (0.4)

6. Secondary Outcome: Mean Sensed Glucose
Description: Assess the mean Dexcom G6 reported sensor glucose values using values uploaded to Dexcom Clarity.The mean sensed glucose was averaged across days 1-7.
Time Frame: Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
mg/dl | 168.4 (28.7) | 177.7 (14.5) | 166.4 (25.7)

7. Secondary Outcome: Percent of Time With Sensed Glucose Less Than 54 mg/dl
Description: Assess the percent of time that the Dexcom G6 reported sensor glucose values less than 54 mg/dl using values uploaded to Dexcom Clarity.The percent of time with sensed glucose less then 54 mg/dl was averaged across days 22-28.
Time Frame: Days 22-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
percentage of time | 0.7 (0.8) | 0.5 (1.1) | 0.8 (1.2)

8. Secondary Outcome: Mean Sensed Glucose
Description: Assess the mean Dexcom G6 reported sensor glucose values using values uploaded to Dexcom Clarity.The mean sensed glucose was averaged across days 22-28.
Time Frame: Days 22-28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
Number analyzed (Participants) | 8 | 8 | 8
mg/dl | 174.0 (22.1) | 184.1 (25.2) | 183.0 (33.1)

ADVERSE EVENTS:
Time Frame: 28 days
Description: All participants that started a visit are included in the adverse events. All subjects completed all visits except one. That subject only completed the start up visit.
Arm/Group | Aerobic Exercise | Anaerobic Exercise | High Intensity Interval Exercise
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=8) | Anaerobic Exercise (N=8) | High Intensity Interval Exercise (N=9)
Shoulder injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Work-related muscle injury
redness and swelling at sensor site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
lightheadedness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
OHSU shall submit for Dexcom's review and comment all publications which result from this Trial. Written copies of results shall be submitted to the Dexcom no later than 45 days before publication and Dexcom shall provide its comments within 30 days, which OHSU will incorporate and honor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT03443713/Prot_SAP_000.pdf